CLINICAL TRIAL: NCT06587087
Title: A Proof of Concept (PoC), Randomized, Controlled Study to Validate the Algorithm and Evaluate the Accuracy, Safety and Pain Level of the Smartest-AE in Comparison to Self-measure Blood Glucose Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Smartest Technologies (Industry)
Collaborators: Israel Innovation Authority (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: SMT000018
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus; Gestational Diabetes Mellitus (GDM); Pre Diabetes
Keywords: Diabetes; Gestational Diabetes Mellitus (GDM); Pre-Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Glucose level device- Smartest-AE (Experimental): The Smartest's System is intended to measure blood glucose levels in home environment. The Smartest's System consists of a disposable single-use device and a mobile app.
  Interventions: Device: Smartest-AE: The lancet that will be used will be the Vitrex Soft Lite lll 28G.
- Commercial Glucometer (Active Comparator)
  Interventions: Device: Smartest-AE: The lancet that will be used will be the Vitrex Soft Lite lll 28G.

INTERVENTIONS:
Device: Smartest-AE: The lancet that will be used will be the Vitrex Soft Lite lll 28G. — The lancet that will be used for all subjects will be the Vitrex Soft Lite lll 28G.

SUMMARY:
The study is conducted in Israel so plain language for the study is exist in Hebrew only

DETAILED DESCRIPTION:
Protocol Title:

A Proof of Concept (PoC), Randomized, Controlled study to validate the algorithm and evaluate the accuracy, safety and pain level of the Smartest-AE in comparison to self-measure Blood Glucose Levels

Investigational Device:

The Smartest-AE

Device Description:

The Smartest's System is intended to measure blood glucose levels in home environment. The Smartest's System consists of a disposable single-use device and a mobile app.

At this study Smartest-AE ("Smartest-AE") will be tested.

Study Overview:

The subjects will be enrolled from the Diabetes Mellitus (DM) clinics in the hospitals, endocrinological clinic, Internal divisions, obstetrics and gynecology department, diabetes in pregnancy and maternal and fetal medicine clinics.

Study subjects will be consecutively screened and enrolled into the study. The study will include up to 300 subjects, men and women aged 18 to 80.

The trial will encompass two distinct populations:

Group 1- Diabetes Mellitus Patients At least 100 subjects who diagnosed with Type I/Type II DM or GDM (Gestational Diabetes Mellitus), who regularly prick their fingers to monitor blood glucose levels and willing to participate in the study, and

Group 2- High risk individuals. at least 100 individuals who do not typically engage in finger pricking but are at high risk of developing prediabetes or diabetes due to to one of the following various risk factors:

* BMI > 25
* Age 45 or older
* Have a parent or sibling with type 2 diabetes
* Have ever had gestational diabetes
* Hypercholesterolemia - according to blood level and\or using medication for lowering cholesterol
* Dyslipidemia - according to blood level and\or using medication for lowering lipids Or any other risk factor according to the staff's discretion.

The study will be conducted in 2 stages:

Stage I- Algorithm verification- Blood glucose levels will be taken from the first 30 subjects in order to verify the algorithm. At the end of the enrollment of the first 30 cases an analysis will be done by Smartest's R&D. If the algorithm yields correlation of R2>0.9, based on the calibration curves, the study will proceed to the second phase. In case the calibration does not show the expected R2 the Smartest's R&D will re-assess the algorithm. If correction/ modification to the algorithm will be implemented another 30 subjects will be enrolled to verify the updated algorithm.

If the analysis following algorithm update, yields satisfying results (R2>0.9), the study will proceed to the second stage and the results of the 30 subjects used for verification will be included in the final analysis. If not, the study will be temporarily paused and the device algorithm will be re-assessed by Smartest's R&D for accuracy and precision. Following that, another 30 subjects will be enrolled for algorithm verification. If the expected R2 is not obtained the study will be terminated.

Blood glucose levels will be measured for all 30/60/90 subjects using 2 devices:

1. The Smartest-AE blood sample analyzer and
2. A commercial standard reference approved glucometer including approved needles and strips.

The lancet that will be used for all subjects will be the Vitrex Soft Lite lll 28G.

All Subjects will complete a Numeric Rating Scale (NRS) questionnaire (Appendix A) to determine their level of pain from each device. NRS will be completed following each finger's pricking

Following NRS completion, blood will be taken from the subject's veins for blood glucose level that will be measured by the site's local lab.

NRS will not be completed following blood taken from the vein.

Stage II- Following algorithm verification and Smartest's approval to continue to stage II at least 200 subjects will be recruited.

Blood Glucose levels will be taken from each subject using the 2 devices; the Smartest-AE and the commercial glucometer.

The blood levels' results of the Smartest-AE will be compared to the commercial approved glucometer in order to assess accuracy. Subjects' comfort/pain level will be assessed following each finger's pricking using the Numeric Rating Scale (NRS) questionnaire

All Subjects will complete the NRS questionnaire to determine their level of pain from each device.

Following NRS completion, blood will be taken from the subject's veins for blood glucose level that will be measured by the site's local lab.

NRS will not be completed following blood taken from the vein. No follow-up period is expected.

Fingers III (middle) and IV (ring) of the non-dominant hand, will be pricked. Randomization will be used to allocate subjects that will be first tested with the Smartest-AE device and subjects that will be first tested with the commercial device. Finger III will always be the first to be pricked.

It was decided that subject IDs' even numbers will have the first prick with the Smartest-AE and subject IDs' odd numbers will have the first prick with the commercial device at each of the groups (1 and 2).

In case the device shows 'error 'or the results seems objectively, to be unreasonable (for eg: extremely high or low blood glucose level result that does not reflect subject physical condition at the time of test), another attempt will be done to achieve the blood glucose level. If the error will be obtained in the first test, then NRS will be completed by the subject subsequently to the test and the second attempt will be done only after the second (reference device) test will be performed. Up to 2 attempts are allowed for each system. Subject that has measurement results only from one system will be excluded from the analysis.

In case failings will be occurred in the venous blood test (either during the blood taking (problematic veins, etc.) or error received from the lab (hemolytic blood, etc.)), a second attempt will not be done and the result will be indicated as missing.

Study Population:

Adults volunteers, men and women, at least 25% of each gender at each group, at the ages of 18- 80 years old, diagnosed with Type I/Type II DM or GDM (Gestational diabetes Mellitus), who regularly prick their fingers to monitor blood glucose levels (Group 1, Diabetes Mellitus patients) and High risk individuals who do not typically engage in finger pricking but are at high risk of developing prediabetes or diabetes due to various risk factors (Group 2).

Hospital personnel are allowed to participate in this study as long they are not subjected directly to the principal investigator.

All subjects will confirm their willingness to participate in the study by signing an Informed Consent Form (ICF).

Study Objective:

To validate the algorithm and to evaluate the accuracy, safety and pain level of the Smartest-AE

Inclusion Criteria:

1. Man or Woman, 18 through 80 years of age
2. Diagnosed with either:

   * Group 1: Type I/II Diabetes Melitus/ GDM who regularly prick his/her fingers to monitor blood glucose levels or,
   * Group 2: High risk individuals who do not typically engage in finger pricking but are at high risk of developing prediabetes or diabetes due to one of the following various risk factors:

     * BMI > 25
     * Age 45 or older
     * Have a parent or sibling with type 2 diabetes
     * Have ever had gestational diabetes
     * Hypercholesterolemia - according to blood level and\or using medication for lowering cholesterol
     * Dyslipidemia- according to blood level and\or using medication for lowering lipids
     * Or any other risk factor according to the staff's discretion
3. Able to self-test using a glucose level device
4. Subject is willing and able to comply with protocol requirements and has provided a signed informed consent form (ICF)

Exclusion Criteria:

1. Subject suffers from neuropathy, chronic pains, pain diseases, impaired sensation in the fingers' area
2. Subject diagnosed with dementia
3. Subject diagnosed with major psychiatric disorders
4. Subject use Narcotics or Analgesics, chronically or at the time of enrollment to the study and up to 4 hours prior to first test of the study
5. Any other medical condition that is considered not eligible by the medical team members
6. Subject Is not capable to report pain levels, objectively
7. Participation in an interventional study at the time of enrollment to this study.

Study Duration :

One year depending on rate of subject recruitment. Duration for each participant: A single visit for couple of hours in the clinic or at the department during hospitalization.

Primary Endpoints:

Stage I- Smartest-AE system algorithm verification (R2>0.9) Stage II- Assess the accuracy of the Smartest-AE glucose measurements' results in comparison to the results received from a commercial approved glucometer.

Secondary Efficacy Endpoints:

1. Subjects' pain level of the Smartest-AE vs. the commercial lancet using the NRS questionnaire
2. Assess the accuracy of the Smartest-AE glucose measurements' results and the commercial glucometer results in comparison to the blood glucose level results of the venous blood test received from the local site's lab

Safety Endpoint:

Any adverse events reported throughout the study following finger pricking will be recorded, including severity (Adverse events such as: infection, exceptional bleeding, blisters, etc.)

Sample size:

The sample size was calculated based on the expected correlation between the commercial glucometer and the Smartest-AE using the G*Power software (version 3.1.9.6), focusing on the Pearson correlation coefficient. The following parameters were used:

Test Type: Exact, Correlation: Bivariate normal model. Tail(s): Two-tailed test. Effect Size (ρ H1): A correlation coefficient of 0.3, reflecting a realistic expectation of the correlation between the variables.

α Error Probability: The alpha level was set at 0.05, maintaining the standard criterion for statistical significance, where there is a 5% chance of a Type I error.

Power (1-β Error Probability): The power was set at 80% (0.8), indicating that there is an 80% probability of correctly rejecting the null hypothesis when it is false.

Correlation ρ H0: The null hypothesis correlation was set to 0, assuming no correlation between the variables.

The calculation results yielded a total sample size of 84 samples.

Smartest company received a grant from the Israel Innovation Authority (IIA). As part of the grant the IIA set a milestone of conducting a clinical trial in 200 subjects for this study purposes. Therefore, the study population size is higher than the necessary sample size.

Statistical Analysis:

Descriptive Statistics: Data will be described by group using mean, standard deviations, median, minimum, and maximum for continuous variables, and counts and proportions for categorical variables.

Subgroup Analysis Stratification by Experience: Differences in reported pain levels between experienced (Group 1) and naïve (Group 2) subjects will be tested using a regression analysis.

Gender Analysis: Differences in reported pain levels will be tested across gender, ensuring at least 25% representation from each gender in both groups.

Software and Data Management Software: All statistical analyses will be conducted using R software. R packages such as "ggplot2" for data visualization and "dplyr" for data manipulation will be utilized to handle and analyze the study data.

Data Management: Data will be coded and stored securely with access restricted to authorized personnel only.

Tables and Figures Table 1: Demographic and Baseline Characteristics by Group. Table 2: Summary Statistics of Blood Glucose Measurements from Smartest-AE, Commercial Glucometer, and Blood Tests.

Table 3: Subgroup Analysis of Pain Levels. Figure 1: correlation plot of Blood Glucose Measurements from Smartest-AE, Commercial Glucometer, and Blood Tests.

Figure 2: Raincloud plots of Pain Levels Reported on NRS by gender.

Handling of Missing Data Missing Data Policy: Subjects missing measurements from either the Smartest-AE or the commercial glucometer will be excluded from the analysis.

Data Imputation: No imputation will be performed for missing glucose measurements; only complete case analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Man or Woman, 18 through 80 years of age
2. Diagnosed with either:

   * Group 1: Type I/II Diabetes Melitus/ GDM who regularly prick his/her fingers to monitor blood glucose levels or,
   * Group 2: High risk individuals who do not typically engage in finger pricking but are at high risk of developing prediabetes or diabetes due to one of the following various risk factors:

     * BMI > 25
     * Age 45 or older
     * Have a parent or sibling with type 2 diabetes
     * Have ever had gestational diabetes
     * Hypercholesterolemia - according to blood level and\or using medication for lowering cholesterol
     * Dyslipidemia- according to blood level and\or using medication for lowering lipids
     * Or any other risk factor according to the staff's discretion
3. Able to self-test using a glucose level device
4. Subject is willing and able to comply with protocol requirements and has provided a signed informed consent form (ICF)

Exclusion Criteria:

* 1. Subject suffers from neuropathy, chronic pains, pain diseases, impaired sensation in the fingers' area 2. Subject diagnosed with dementia 3. Subject diagnosed with major psychiatric disorders 4. Subject use Narcotics or Analgesics, chronically or at the time of enrollment to the study and up to 4 hours prior to first test of the study 5. Any other medical condition that is considered not eligible by the medical team members 6. Subject Is not capable to report pain levels, objectively 7. Participation in an interventional study at the time of enrollment to this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Algorithm verification | 1 months
  Stage I- Smartest-AE system algorithm verification (R2>0.9)
Stage II- Accuracy | 3 months
  Stage II- Assess the accuracy of the Smartest-AE glucose measurements' results in comparison to the results received from a commercial approved glucometer.

SECONDARY OUTCOMES:
Pain Level | 4 months
  Subjects' pain level of the Smartest-AE vs. the commercial lancet using the NRS questionnaire
accuracy vs. lab results | 4 months
  Assess the accuracy of the Smartest-AE glucose measurements' results and the commercial glucometer results in comparison to the blood glucose level results of the venous blood test received from the local site's lab

OTHER OUTCOMES:
Safety | 4 months
  Any adverse events reported throughout the study following finger pricking will be recorded, including severity (Adverse events such as: infection, exceptional bleeding, blisters, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Enav Yefet, MD, Principal Investigator — Baruch Padeh Medical center Poriya
Locations (1):
- The BARUCH PADEH Medical Center, Poriya, Poria – Neve Oved, The Lower Galilee, Israel

IPD SHARING:
Plan to Share IPD: Undecided